CLINICAL TRIAL: NCT06434389
Title: A Point-of-care Electrochemical-based Device for Rapid Detection of Fibrinogen on Type A Aortic Dissection Surgery
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0561
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-02

CONDITIONS: Hypofibrinogenemia
MeSH Terms: conditions — Afibrinogenemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The patients undergoing routine coagulation tests: Part1 Phase I-Laboratory calibration. Phase II-Assay performance using clinical samples. using human biological samples already collected for routine coagulation analysis.
  Part2 Subject underwent surgery for acute type A aortic dissection and requires routine TEG test， residual blood samples collected for fibrinogen detection by the Clauss method and electrochemical method.
  Interventions: Diagnostic Test: the Electrochemical-based device

INTERVENTIONS:
Diagnostic Test: the Electrochemical-based device — Electrochemical-based device for rapid detection of fibrinogen is a novel POC diagnostic method, which is suitable for operating theatres and emergency rooms.

SUMMARY:
This study compares the results of the existing fibrinogen concentration monitoring technology to the Electrochemical-based device, a point-of-care and rapid method,using a small amount of extra blood obtained in Type A Aortic Dissection Surgery.

DETAILED DESCRIPTION:
Electrochemical-based device for rapid detection of fibrinogen is a novel POC diagnostic method, which is suitable for operating theatres and emergency rooms.

The novel fibrinogen detection based on Gel electrodes combined with immunobiosensing strategies and use magnitude of current to characterize the fibrinogen concentration , which will be a POC assay of fibrinogen detection for critically ill patients.

This single-center, prospective, observational pilot study will evaluate the analytical performance as well as compared to conventional Clauss laboratory reference method.

ELIGIBILITY:
Part1 Phase I-Laboratory calibration. The electrochemical method was employed to detect the fibrinogen concentration of standard quality control materials with varying concentration gradients, and the corresponding current values were recorded for constructing a standard curve of fibrinogen concentration.

Phase II-Assay performance using clinical samples. Subject is 18 years and underwent routine hemostasis analysis. using human biological samples already collected for routine hemostasis analysis, The samples were centrifuged at 2500g for 15 min at room temperature, to obtain PPP (residual platelet count of <10 × 10^9/L) and stored at-20℃used for determination by electrochemical method within 2 weeks, Each clinical sample was tested three times

Part2

Inclusion Criteria:

Subject underwent surgery for acute type A aortic dissection at our hospital, Subject is 18 years, Subject requires routine TEG measurement, Subject use human fibrinogen concentrate during surgery.

Exclusion Criteria:

Use Extracorporeal Membrane Oxygenation after surgery, inability to obtain written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited at the Second Affiliated Hospital Zhejiang University School of Medicine. For part 1:The study participants will be adult underwent routine hemostasis analysis. For part 2:The study participants will be adult underwent surgery for acute type A aortic dissection and requires routine TEG test, residual blood samples collected for fibrinogen detection by the Clauss method and electrochemical method.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The fibrinogen concentration values obtained using the Clauss method and electrochemical method were compared | 1 day

SECONDARY OUTCOMES:
the time of the two detection methods | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No